CLINICAL TRIAL: NCT00034866
Title: Double-Blind, Randomized, Dose Optimization Trial of Three Doses of Tipranavir Boosted With Low Dose Ritonavir (TPV/RTV) in Multiple Antiretroviral Drug-Experienced Subjects.
Brief Title: Dose Ranging Trial of Tipranavir/Ritonavir in Treatment-Experienced HIV Infected Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BI 1182.52
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV; treatment experienced; Boehringer; tipranavir; ritonavir
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Protease inhibitor tipranavir

SUMMARY:
The purpose of this research study is to determine which of three different dose combinations of tipranavir and ritonavir, when taken with a standard approved anti-HIV drug therapy, is most effective and safe. Tipranavir is an investigational protease inhibitor which has been demonstrated to have in vitro activity against HIV-1.

DETAILED DESCRIPTION:
This study will be conducted in HIV+, multiple ARV medication experienced patients. All patients must have received treatment from each of three ARV classes: NRTIs, NNRTIs and PIs, have received at least two PI-based ARV regimens (may include the current regimen) with a viral load greater than or equal to 1000 copies/mL at the time of study entry. The two separate PI-based regimens must each have been taken for at least 3 months. At least one resistance-conferring PI-mutation (from a pre-established panel) must be present. Baseline genotypic screening will be performed and will be used in conjunction with ARV medication history to determine new background therapy for each individual subject to use.

Following genotypic screening at baseline, qualifying subjects will be randomized to one of three blinded treatment regimens. Subjects will discontinue their current protease inhibitor and initiate TPV/RTV for 2 weeks of functional monotherapy. Thereafter, the background ARV medications will be optimized and subjects will remain on blinded TPV/RTV plus optimized background therapy for the duration of the trial. Trial duration ranges between 12-32 weeks, depending on when the subject is entered into the trial and the interim analyses for determination of optimized TPV/RTV regimen is completed. On determination of the optimal TPV/RTV dose, subjects may opt to continue open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to trial participation.
2. HIV-1 infected males or females >= 18 years of age.
3. At least 3 months experience taking NRTIs, NNRTI(s), and PIs.
4. Current PI-based ARV medication regimen for at least 3 months prior to randomization, and at least 3 months experience taking at least one other PI-based regimen.
5. HIV-1 viral load >= 1000 copies/mL at screening.
6. Genotypic resistance report indicating one or more primary PI resistance mutation(s), including 30N, 46I/L, 48V, 50V, 82A/F/T, 84V or 90M, with not more than one of 82 A/F/T or 84V or 90M.
7. Acceptable screening laboratory values that indicate adequate baseline organ function. Laboratory values are considered to be acceptable if severity is no higher than Grade 3 GGT, Grade 2 cholesterol or triglycerides, and no higher than Grade 1 for all other tests based on the DAIDS Grading Scale. All laboratory values outside these limits are subject to approval by BI.
8. Acceptable medical history, as assessed by the investigator, with chest X-ray and ECG within 1 year of study participation.
9. Willingness to abstain from ingesting substances which may alter plasma study drug levels by interaction with the cytochrome P450 system, such as: grapefruit or Seville oranges or their products; herbal preparations containing St. John's Wort or milk thistle, and garlic supplements.
10. A prior AIDS defining event is acceptable as long as it has resolved or the subject has been on stable treatment for at least 2 months.

Exclusion Criteria:

1. ARV medication naïve.
2. Female subjects who:

   * have a positive serum pregnancy test at screening or during the study
   * are breast feeding
   * are planning to become pregnant
   * are not willing to use two barrier methods of contraception (e.g. latex condom plus spermicidal jelly/foam).
3. Any active opportunistic infection within 60 days before study entry.
4. Active Hepatitis B or C disease defined as HBsAg positive or HCV RNA positive with AST/ALT >Grade 1.
5. Prior tipranavir use.
6. Use of investigational medications within 30 days before study entry or during the trial. Some expanded access drugs may be acceptable; must be approved by BI. Tenofovir, investigational at time of preparation of this protocol, is acceptable.
7. Use of concomitant drugs which may significantly reduce plasma levels of the study medications.
8. Use of immunomodulatory drugs (e.g. interferon, cyclosporin, hydroxyurea, interleukin-2).
9. Active substance abuse.
10. Inability to swallow TPV or RTV capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2002-04; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Locations (51):
- United States (50):
  - Phoenix Body Positive, Phoenix, Arizona
  - Orange County Center for Special Immunology, Fountain Valley, California
  - Living Hope Clinical Trials Inc., Long Beach, California
  - AHF Research Center, Los Angeles, California
  - University of So. California / LA County USC Medical Center, Los Angeles, California
  - ID Care, Inc., Los Angeles, California
  - Tower I.D. Medical Assoc., Inc., Los Angeles, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - University of California San Francisco Positive Health Program Research, San Francisco, California
  - Pacific Horizon Medial Group, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - (IDC) Research Institute, Altamonte Springs, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Jackson Medical Tower, Miami, Florida
  - Steinhart Medical Associates, South Miami, Florida
  - Hillsborough County Health Dept., Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta VA Medical Center, Dept. of ID, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - CORE Center, Cook County Hospital, Chicago, Illinois
  - Rush Presbyterian/St. Luke's Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - HIV Outpatient Program (H.O.P.), New Orleans, Louisiana
  - John's Hopkins University School of Medicine, Baltimore, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - CRI Community Research Initiative, Springfield, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Hospital, Infectious Diseases Dept., Detroit, Michigan
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - Washington University AIDS Clinical Trial Unit, St Louis, Missouri
  - Wellness Center, Las Vegas, Nevada
  - ID Care, Inc., Hillsborough, New Jersey
  - ID Care, Inc., Randolph Township, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of New York at Stony Brook, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center Infectious Diseases Clinic, Durham, North Carolina
  - Jemsek Clinic, Huntersville, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Infect. Disease Institute, Clinical Trials Unit, Oklahoma City, Oklahoma
  - Burnside Clinic, Columbia, South Carolina
  - Vanderbilt University - AIDS Clinical Trial Unit, Nashville, Tennessee
  - Nelson-Tebedo Clinic, Dallas, Texas
  - Gathe Clinic, Houston, Texas
  - Infectious Disease Physicians Research, Annandale, Virginia
- Clinical Research Puerto Rico, San Juan, Puerto Rico